CLINICAL TRIAL: NCT05532852
Title: Efficacy and Safety Evaluation of Paxlovid for COVID-19: a Real-world Case-control Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Jieming QU, Principal Investigator, Ruijin Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY01004
Record Dates: First submitted 2022-09-06; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: COVID-19 Pneumonia
MeSH Terms: interventions — Standard of Care; nirmatrelvir and ritonavir drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard-of-care (Sham Comparator)
  Interventions: Drug: standard-of-care
- standard-of-care plus Paxlovid (Experimental)
  Interventions: Drug: standard-of-care plus Paxlovid

INTERVENTIONS:
Drug: standard-of-care plus Paxlovid — standard-of-care plus Paxlovid
  Arms: standard-of-care plus Paxlovid
Drug: standard-of-care — standard-of-care
  Arms: standard-of-care

SUMMARY:
COVID-19 is currently one of the serious public health challenges worldwide, and there is a great need to develop effective treatments. Paxlovid is a Pfizer-developed oral new drug for the treatment of COVID-19. Paxlovid, which is used to treat adult patients with mild to moderate COVID-19 who have high-risk factors for progression to severe disease, was conditionally approved for marketing in the United States and China in December 2021 and February 2022, respectively. Clinical trials have shown that this drug can significantly reduce the progression from mild to severe disease and the rate of hospitalization and mortality. However, due to the limitations of clinical trials in the subject selection, there is still insufficient knowledge about the efficacy and safety of Paxlovid in a real-world population. Relevant studies on this drug in real-world people, especially in Chinese populations, have not been reported. Therefore, this study was designed to investigate the efficacy and safety of Paxlovid on sufferers of COVID-19 through a retrospective, real-world analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed COVID-19 who had taken more than one dose of Paxlovid.

Exclusion Criteria:

* Age < 18 years-old;
* Pregnancy;
* Data missing > 20%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 728 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | 28 days since the diagnosis of COVID-19
  the mortality of the subjects within 28 days since the diagnosis of COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Jieming Qu, Principal Investigator — Rui-jin Hospital, Shanghai Jiao-tong University School of Medicine, Shanghai,
Locations (1):
- Ruijin Hospital, Medical School of Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No